CLINICAL TRIAL: NCT01079442
Title: Does Coffee Intake Reduce Postoperative Ileus After Elective Colectomy?
Brief Title: Coffee Trial - Does Coffee Intake Reduce Postoperative Ileus After Elective Colectomy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Nuh Rahbari, chief resident, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NNR-6
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Colectomy
Keywords: postoperative ileus after colonic resections
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment arm: coffee (Active Comparator): coffee administration
  Interventions: Other: Postoperative coffee
- Water arm (Placebo Comparator): The control drink consists of 100 ml warm water
  Interventions: Other: water

INTERVENTIONS:
Other: Postoperative coffee — schedule for coffee administration for the present trial was chosen as follows (starting 6 hours postoperatively):
  * 08:00 100mL beverage
  * 12:00 100mL beverage
  * 16:00 100mL beverage
  Other Names: Lavazza Blue Espresso Dolce 100% Arabica coffee
  Arms: Treatment arm: coffee
Other: water — The control drink consists of 100 ml warm water which is administered according a same fixed schedule as Group A starting 6 hours postoperatively:
  * 08:00 100mL beverage
  * 12:00 100mL beverage
  * 16:00 100mL beverage
  Other Names: tap water
  Arms: Water arm

SUMMARY:
The purpose of the investigators study is to investigate the effects of coffee on the return of bowel function and appetite, length of hospital stay, and complications after elective open colectomy in a prospective randomized trial. The primary efficacy endpoint is time to first bowel movement.

DETAILED DESCRIPTION:
Coffee is a popular beverage. Its effects on general well being, central nervous system and cardiovascular system are well known, but there is limited information regarding its effects on gastrointestinal function.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective open or laparoscopic colectomy
* Age equal or greater than 18 years
* Informed consent

Exclusion Criteria:

* Participation in concurrent intervention trials
* Need for a stoma
* Known hypersensitivity or allergy to coffee
* Expected lack of compliance
* Impaired mental state or language problems
* change in surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Time to first bowel movement | patients postoperative in hospital stay (mean 6 days)
  Time from end of surgery until patient's first bowel movement (i.e. passage of stool).

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Salem Krankenhaus, Heidelberg
  - University hospital, Heidelberg
  - Kreiskrankenhaus GRN Sinsheim, Sinsheim

REFERENCES:
- [Derived] Muller SA, Rahbari NN, Schneider F, Warschkow R, Simon T, von Frankenberg M, Bork U, Weitz J, Schmied BM, Buchler MW. Randomized clinical trial on the effect of coffee on postoperative ileus following elective colectomy. Br J Surg. 2012 Nov;99(11):1530-8. doi: 10.1002/bjs.8885. Epub 2012 Sep 14. PMID 22987303